CLINICAL TRIAL: NCT01569633
Title: Pilot Study for Use of Prokinetics in Early Enteral Feeding of Preterm Infants ; Double Blind; Cross Over Study Comparing Eryththromycin, Metoclopramide and Placebo
Brief Title: Use of Prokinetics in Early Enteral Feeding in Preterm Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: very poor enrollment
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Darshan Shah, M.D., Asst. Professor of Pediatrics, East Tennessee State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ft2011ep
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Feeding Disorder; Nutrition Disorder; Infant,Premature
MeSH Terms: conditions — Feeding and Eating Disorders; Nutrition Disorders; Premature Birth | interventions — Metoclopramide; Erythromycin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): This group of infant will not receive any medication but sugar water or placebo
  Interventions: Drug: placebo
- Metclopramide (Active Comparator): This group of infants will receive Metoclopramide at 0.1mg/kg q8 hrs.
  Interventions: Drug: Metclopramide
- Erythromycin (Active Comparator): mediaction used to treat feeding disorder
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Metclopramide — Dose of metoclopramide is 0.1miligram per kilogram every eight hours for 7-14 days.
  Other Names: reglan
  Arms: Metclopramide
Drug: Erythromycin — Dose of erythromycin is 1 miligram per kilogram every eight hours
  Arms: Erythromycin
Drug: placebo — The dose of sugar water is 1 ml per 8 hours.
  Arms: Placebo

SUMMARY:
Objective of this study are:

1) To determine if medication help extreme preterm infants to tolerate feeding better by reaching full feeding earlier.2) Out of two medication; which one is better for efficacy 1) Erythromycin 2) Metoclopramide. Infants who meet inclusion criteria would be entered to study after parental consent. Infant would be blinded to care givers. Infants will be randomized to receive one of three medication for 7-14 days. If infants fail on one medication they will be allowed to crossover to other medication. Infant would be allowed to treat like other infants. Blindness can be broken if deem necessary by attending neonatologist.

DETAILED DESCRIPTION:
Inclusion Critera:

1. Weight below 1250 grams
2. Age less than 14 days
3. Feeding intolerance; If feeding residual more than 30% on q3 hr feeding; 5 times out of 8 times, feeding residual more than 20% on q4 hr feeding 4 feeding out of 6 feeding or failure to advance feeding of more than 20ml/kg in 72 hrs.

Exclusion Criteria

1. GI malformation or perforation
2. Genetic disorder
3. Parents can't read English. After consent, if infants meet inclusion criteria, he would be allowed to receive one of the following three medication. 1) Erythromycin at 1mg/kg/dose q8 hr 2) Metoclopramide 0.1mg/kg/dose q8 hrs and Placebo. If infant fails to get better, he would be crossover to one of the remaining two.

ELIGIBILITY:
Inclusion Criteria:

1. Weight below 1250 grams
2. Age less than 14 days
3. Feeding intolerance; If feeding residual more than 30% on q3 hr feeding; 5 times out of 8 times, feeding residual more than 20% on q4 hr feeding 4 feeding out of 6 feeding or failure to advance feeding of more than 20ml/kg in 72 hrs.

Exclusion Criteria

1. GI malformation or perforation
2. Genetic disorder
3. Parents can't read English. After consent, if infants meet inclusion criteria, he would be allowed to receive one of the following three medication. 1) Erythromycin at 1mg/kg/dose q8 hr 2) Metoclopramide 0.1mg/kg/dose q8 hrs and Placebo. If infant fails to get better, he would be crossover to one of the remaining two.

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Prokinetics and PLACEBO IN EARLY ENTERAL NUTRITION OF EXTREME PRETERM INFANTS; DOUBLE BLIND CROSS OVER TRIAL | 24 MONTHS
  Time to reach full enteral feeding in both infants. Which of the two medication help better in reaching full enteral feeding.

SECONDARY OUTCOMES:
Comaparison of Prokintics and Placebo in Early Enteral Nutrition of Extreme Preterm Infants; Double blind cross over trial. | 24 months
  Duration of Total Parental Nutrition; duration of direct hyperbilirubinemia,

CONTACTS AND LOCATIONS:
Overall Officials: Darshan S Shah, MD, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States